CLINICAL TRIAL: NCT02386657
Title: Single-center Prospective Evaluation of Sickle Cell Patient Care in the CHU Brugmann Emergency Department
Status: Completed | Type: Observational
Sponsor: Brugmann University Hospital (Other)
Responsible Party: Principal Investigator, Andre Efira, Head of Clinic, Brugmann University Hospital
Other Study IDs: CHUB-Edu
Record Dates: First submitted 2015-03-03; First posted 2015-03-12 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Sickle Cell Disease
Keywords: Sickle Cell Disease; Vaso-occlusive crisis; Emergency management
MeSH Terms: conditions — Anemia, Sickle Cell; Vaso-Occlusive Crises | interventions — Physician Engagement; Pain Management

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Emergency admitted sickle cell disease patients: Sickle Cell Disease Patients admitted inside the Emergency Department of the Brugmann Hospital for a vaso-occlusive crisis.
  Interventions: Other: Satisfaction; Other: Biological parameters; Other: Pain management

INTERVENTIONS:
Other: Satisfaction — Satisfaction questionnaire to be filled in
Other: Biological parameters — Measure of standard routine biological parameters (Hb, GB, Plaq, LDH, CRP, TCA, INR, D Dimers) and dosage of nitrous albumin (PNA).
Other: Pain management — Validated pain scale questionnaire to be filled in

SUMMARY:
Sickle Cell Disease is a serious disease that is life-threatening for patients being homozygous for the SS form or heterozygous for the SC or bthal forms. The CHU Brugmann hospital currently regularly treats about 70 homozygous adult patients and this number is in constant augmentation. The age average of the patients is below 30. The hospital developed a close collaboration with the Queen Fabiola Kids University Hospital to optimize the transition of young sickle cell patients from the pediatric to the adult network.

The emergency care of sickle cell patients remains a source of worry. Even with a correct treatment (Hydroxy-urea or exsanguineous transfusions), patients suffer from frequent sickle cell disease crisis when stress or infection cause hemolysis. The pain level is intolerable and causes emergency hospital admission (2 to 3 crisis per patient per year on average). The crisis are more frequent with poor compliance to the treatments.

There are several obstacles to the rapid and optimal management of these patients:

* fear of causing addiction to heavy pain releaf products (high dosis of morphine)
* lack of biological parameters for the determination of the crisis severity.

The prognostic value of the lactate dehydrogenase (LDH) level in a vaso-occlusive crisis was recently stressed while activation of the coagulation, translated by the elevation of various parameters including the rate of DD dimers, seemed associated with clinical complications. The deleterious role of increased oxidative stress has also been recently demonstrated in patients with sickle cell disease, opening new therapeutic avenues.

This study aims to prospectively evaluate the management of sickle cell patients being admitted in the emergency department for a vaso-occlusive crisis. The level of satisfaction of the patients will be measured.

The investigators will also evaluate the predictive value of several routine biological parameters regarding the severity of the crisis, including the values of nitrous albumin (PNA) as marker of oxydative stress. This last dosage will be made in collaboration with the team of Dr Wayenberg and Pr Bottari in Grenoble.

ELIGIBILITY:
Inclusion Criteria:

* Any sickle cell disease patient being admitted inside the Emergency Department of the Brugmann Hospital for a vaso-occlusive crisis, having signed the informed consent form and being able to fill in the analogic visual questionnaire (EVA).

Exclusion Criteria:

* Patients not being able to sign the informed consent form or fill in the analogic visual questionnaire (EVA)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sickle Cell Disease patients, entering the Emergency Department of the Brugmann Hospital for a vaso-occlusive crisis.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2012-11; Primary Completion 2015-02 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
EVA pain scale | 48 hours
  The pain will be evaluated using the EVA scale (Visual Analogic scale) by the patient himself and by the nursing staff (hetero-anamnesis). Time frames will be: at admission within the emergency department, 1 hour after admission, 3h after admission, 6 hours after admission and, if the pain did not disappear by then, every 6 hours until the pain disappears.

SECONDARY OUTCOMES:
Satisfaction questionnaire | 10 days
  Satisfaction of the patient regarding the management of his/her pain management.
Morphine amount | 10 days
  Morphine amount administrated within the Emergency Department and during hospitalization length.
Hospitalisation length | 10 days
  Time needed being hospitalized in order to control the pain level after the initial episode.
Standard biological parameters | at hospital emergency service admission
  Dosage of the standard biological parameters (Hb, GB, Plaq, LDH, CRP, TCA, INR, D Dimers) and the nitrous albumin levels (PNA) at hospital admission.
Standard biological parameters | 10 days
  Dosage of the standard biological parameters (Hb, GB, Plaq, LDH, CRP, TCA, INR, D Dimers) and the nitrous albumin levels (PNA) at the end of hospitalisation.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Agnès Azerad, MD, Principal Investigator — CHU Brugmann
Locations (1):
- CHU Brugmann, Brussels, Belgium

REFERENCES:
- [Background] Platt OS, Thorington BD, Brambilla DJ, Milner PF, Rosse WF, Vichinsky E, Kinney TR. Pain in sickle cell disease. Rates and risk factors. N Engl J Med. 1991 Jul 4;325(1):11-6. doi: 10.1056/NEJM199107043250103. PMID 1710777
- [Background] Solomon LR. Treatment and prevention of pain due to vaso-occlusive crises in adults with sickle cell disease: an educational void. Blood. 2008 Feb 1;111(3):997-1003. doi: 10.1182/blood-2007-07-089144. Epub 2007 Oct 16. PMID 17940207
- [Background] Brookoff D, Polomano R. Treating sickle cell pain like cancer pain. Ann Intern Med. 1992 Mar 1;116(5):364-8. doi: 10.7326/0003-4819-116-5-364. PMID 1736768
- [Background] Payne R. Sickle cell anemia and pain: will data prevail over beliefs? Ann Emerg Med. 2009 May;53(5):596-7. doi: 10.1016/j.annemergmed.2008.10.022. No abstract available. PMID 19380037
- [Background] Zempsky WT. Treatment of sickle cell pain: fostering trust and justice. JAMA. 2009 Dec 9;302(22):2479-80. doi: 10.1001/jama.2009.1811. No abstract available. PMID 19996405
- [Background] Tanabe P, Artz N, Mark Courtney D, Martinovich Z, Weiss KB, Zvirbulis E, Hafner JW. Adult emergency department patients with sickle cell pain crisis: a learning collaborative model to improve analgesic management. Acad Emerg Med. 2010 Apr;17(4):399-407. doi: 10.1111/j.1553-2712.2010.00693.x. PMID 20370779
- [Background] Tanabe P, Hafner JW, Martinovich Z, Artz N. Adult emergency department patients with sickle cell pain crisis: results from a quality improvement learning collaborative model to improve analgesic management. Acad Emerg Med. 2012 Apr;19(4):430-8. doi: 10.1111/j.1553-2712.2012.01330.x. PMID 22506947
- [Background] Anie KA, Grocott H, White L, Dzingina M, Rogers G, Cho G. Patient self-assessment of hospital pain, mood and health-related quality of life in adults with sickle cell disease. BMJ Open. 2012 Jul 2;2(4):e001274. doi: 10.1136/bmjopen-2012-001274. Print 2012. PMID 22761289
- [Background] Stankovic Stojanovic K, Steichen O, Lefevre G, Bachmeyer C, Avellino V, Grateau G, Girot R, Lionnet F. High lactate dehydrogenase levels at admission for painful vaso-occlusive crisis is associated with severe outcome in adult SCD patients. Clin Biochem. 2012 Dec;45(18):1578-82. doi: 10.1016/j.clinbiochem.2012.07.114. Epub 2012 Aug 8. PMID 22892192
- [Background] Ataga KI, Brittain JE, Desai P, May R, Jones S, Delaney J, Strayhorn D, Hinderliter A, Key NS. Association of coagulation activation with clinical complications in sickle cell disease. PLoS One. 2012;7(1):e29786. doi: 10.1371/journal.pone.0029786. Epub 2012 Jan 11. PMID 22253781
- [Background] Rees DC, Gibson JS. Biomarkers in sickle cell disease. Br J Haematol. 2012 Feb;156(4):433-45. doi: 10.1111/j.1365-2141.2011.08961.x. Epub 2011 Nov 28. PMID 22122125
- [Background] Schnog JB, Teerlink T, van der Dijs FP, Duits AJ, Muskiet FA; CURAMA Study Group. Plasma levels of asymmetric dimethylarginine (ADMA), an endogenous nitric oxide synthase inhibitor, are elevated in sickle cell disease. Ann Hematol. 2005 May;84(5):282-6. doi: 10.1007/s00277-004-0983-3. Epub 2004 Dec 14. PMID 15599544
- [Background] Nur E, Brandjes DP, Teerlink T, Otten HM, Oude Elferink RP, Muskiet F, Evers LM, ten Cate H, Biemond BJ, Duits AJ, Schnog JJ; CURAMA study group. N-acetylcysteine reduces oxidative stress in sickle cell patients. Ann Hematol. 2012 Jul;91(7):1097-105. doi: 10.1007/s00277-011-1404-z. Epub 2012 Feb 10. PMID 22318468
- [Background] Wayenberg JL, Ransy V, Vermeylen D, Damis E, Bottari SP. Nitrated plasma albumin as a marker of nitrative stress and neonatal encephalopathy in perinatal asphyxia. Free Radic Biol Med. 2009 Oct 1;47(7):975-82. doi: 10.1016/j.freeradbiomed.2009.07.003. Epub 2009 Jul 8. PMID 19591921